CLINICAL TRIAL: NCT04496882
Title: The Clinical Efficacy of Tenofovir Alafenamide-switching Therapy in Patients With Chronic Hepatitis B Experiencing Clinical Flare-up After Discontinuation of Nucleos[t]Ide Analogues Therapy
Brief Title: Chronic Hepatitis b Patients Switch to tAf After Discontinuation of Nucleoside Analogue
Acronym: CHANGE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other); Taipei City Hospital (Other Government); Chiayi Christian Hospital (Other); Dalin Tzu Chi General Hospital (Other); E-DA Hospital (Other); Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201911095MIPD
Record Dates: First submitted 2020-07-26; First posted 2020-08-03 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hepatitis b; Hepatitis B Reactivation
Keywords: HBV,clinical relapse,Vemlidy (TAF)
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Switching therapy cohort (Experimental): single arm, open label Patients will receive Vemlidy (tenofovir alafenamide, TAF) 25mg, daily for 48 weeks
  Interventions: Drug: Vemlidy
- Historical continuing therapy cohort (No Intervention): By retrospectively review medical records, The patients continued the original regimen (ETV, TDF) for retreatment (within 3 months of clinical relapse)

INTERVENTIONS:
Drug: Vemlidy — 25mg Tenofovir Alafenamide
  Other Names: Tenofovir Alafenamide (TAF)
  Arms: Switching therapy cohort

SUMMARY:
We will conduct a phase 4, multicenter, open-label trial at 7 academic centers in Taiwan.

Chronic hepatitis B patients receiving oral antiviral therapy (entecavir [ETV], tenofovir disoproxil fumarate [TDF]) for at least 2 years, and fulfil the following nucleos(t)ide analogs discontinuation criteria. After nucleos(t)ide analogs discontinuation, patients had a clinical relapse and retreatment regimen switches to TAF.

The protocol will be approved by Institutional Review Board (IRB) or Research ethic committee (REC) of each site and will be conducted in accordance with the principles of Declaration of Helsinki and the International Conference on Harmonization for Good Clinical Practice. Each patient provides written informed consent before enrollment.

DETAILED DESCRIPTION:
Tenofovir alafenamide (TAF) is a new generation of oral antiviral drugs with similar antiviral activities to tenofovir disoproxil fumarate (TDF) and reduces the adverse effects of nephrotoxicity and bone mineral density reduction. This drug has already been reimbursed by National Health Insurance, and can be used for the treatment of patients with chronic hepatitis B.

This is a single-arm prospective clinical trial to enroll patients who discontinued entecavir (ETV) and tenofovir disoproxil fumarate (TDF) and experienced a clinical hepatitis flare up. They can be retreated with TAF for 48 weeks without postponing a 3-month observation period for alanine aminotransferase (ALT) level. The virological control, ALT level recovery, and changes in liver fibrosis, hepatitis B surface antigen, hepatitis B core-associated antigen, and renal function will be observed during retreatment. In addition, a group of patients with the same characteristics who received retreatment with entecavir or TDF will be collected as a control group for comparison. We believe this study can help us understand the clinical benefits of switching to TAF for retreatment after hepatitis flare in patients to discontinue oral antiviral agents.

ELIGIBILITY:
Inclusion Criteria A. Switching therapy cohort

1. Chronic hepatitis B patients receiving oral antiviral therapy (ETV, TDF) for at least 2 years, and fulfil the following NUCs discontinuation criteria (1)HBeAg-positive patients achieving HBeAg seroclearance, and received at least 1-year consolidation therapy (2) HBeAg-negative patients achieving undetectable HBV DNA for more than 1 year (on 3 occasions, 6 months apart)
2. After NUC discontinuation, patients had a clinical relapse (HBV DNA > 2000 IU/mL, and ALT > 2x ULN)
3. The retreatment regimen switches to TAF (within 3 months of clinical relapse)

B. Historical continuing therapy cohort

1. Chronic hepatitis B patients receiving oral antiviral therapy (ETV, TDF) for at least 2 years, and fulfil the following NUCs discontinuation criteria (1) HBeAg-positive patients achieving HBeAg seroclearance, and received at least 1-year consolidation therapy (2) HBeAg-negative patients achieving undetectable HBV DNA for more than 1 year(on 3 occasions, 6 months apart)
2. After NUC discontinuation, patients had a clinical relapse (HBV DNA > 2000 IU/mL, and ALT > 2x ULN)
3. The patients continued the original regimen (ETV, TDF) for retreatment (within 3 months of clinical relapse)

Exclusion Criteria

1. Patients who do not fulfill the discontinuation criteria
2. Patients who have HCV, HDV or HIV co-infection
3. Patients who discontinue lamivudine, adefovir, or telbivudine therapy
4. Patients with liver cirrhosis by ultrasonography and clinical diagnosis

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of virological remission (HBV DNA <20 IU/mL) | 48 weeks
  We will calculate the rate of virological remission (HBV DNA <20 IU/mL) after retreatment

SECONDARY OUTCOMES:
Rate of ALT normalization (ALT < 40 U/L) after retreatment | 48 weeks
  We will calculate the rate of ALT normalization (ALT < 40 U/L) after retreatment
Rate of HBsAg change after retreatment compared with baseline | 48 weeks
  We will investigate the rate of HBsAg change after retreatment compared with the baseline HBsAg
Rate of HBcrAg change after retreatment compared with baseline | 48 weeks
  We will investigate the rate of hepatitis B core-related antigen (HBcrAg) change after retreatment compared with baseline HBcrAg
Rate of M2BPGi level change after retreatment compared with baseline | 48 weeks
  We will investigate the rate of Mac-2 binding protein glycosylation isomer (M2BPGi) level change after retreatment compared with baseline M2BPGi level

CONTACTS AND LOCATIONS:
Overall Officials: Tung-Hung Su, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (7):
- Taiwan (7):
  - Buddhist Tzu Chi General Hospital, Da-Lin Branch, Chiayi City
  - Chia-Yi Christian Hospital, Chiayi City
  - National Taiwan University Hospital, Yun-Lin branch, Douliu
  - E-da hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Buddhist Tzu-Chi General Hospital Taipei Branch, Taipei
  - Taipei City Hospital, Renai Branch, Taipei

IPD SHARING:
Plan to Share IPD: No